CLINICAL TRIAL: NCT00709683
Title: An Observational Study Evaluating the Safety and Efficacy of the Treatment With Biphasic Insulin Aspart (NovoMix® 30 FlexPen®) in the Treatment of Type 2 Diabetics After Failing on Basal/ Intermediate Mono or Combination Therapy
Brief Title: Observational Study to Evaluate the Safety of NovoMix® 30 FlexPen®
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3572
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: NovoMix® 30

SUMMARY:
This study is conducted in Africa. The aim of this observational study is to evaluate the incidence of adverse events while using NovoMix® 30 FlexPen® under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes having failed on basal insulin with or without OAD
* HbA1c greater than 7.0%

Exclusion Criteria:

* Subjects being unlikely to comply with protocol requirements
* Subjects who previously enrolled in this study
* Subjects with hypersensitivity to biphasic insulin aspart or any of the excipients
* Women who are pregnant, breast feeding and women in child bearing capacity who are not using reliable contraceptive method

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetic patients
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence of major hypoglycaemic events reported as serious adverse drug reactions | during 26 weeks of treatment

SECONDARY OUTCOMES:
Number of serious adverse drug reactions | during 26 weeks of treatment
Number of serious adverse events | during 26 weeks of treatment
Number of all major (daytime and nocturnal) hypoglycaemic events | during 26 weeks of treatment
Number of all minor (daytime and nocturnal) hypoglycaemic events | during 26 weeks of treatment
Weight (BMI) change from baseline | At the end of the study
HbA1c change from baseline | At the end of the study
Percentage of patients reaching the target of HbA1c of less than or equal to 7.0% | At the end of the study
Average (mean) fasting plasma glucose level | At the end of the study
Average post-breakfast (90-120 mins), post-lunch (90-120 mins), post-dinner (90-120 mins) plasma glucose level | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tunisia, Tunisia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com